CLINICAL TRIAL: NCT01626235
Title: Acute Management of Pain From the Emergency Department: A National, Emergency Department-Based Prospective Post-Intervention Registry of Non-Opioid and Opioid Management of Acute Pain
Brief Title: AMPED Outcomes Registry of Post-ED Pain Management
Acronym: AMPED
Status: Completed | Type: Observational
Sponsor: Radnor Registry Research, Inc (Industry)
Collaborators: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RRR-LUIT-01
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Soft Tissue Injuries; Gouty Arthritis; Fractures; Ureteral Colic; Dysmenorrhea
Keywords: pain control; fractures; sprains; strains; dysmenorrhea; kidney stones; gouty arthritis; opioids; NSDAIDs; Emergency Department; patient reported outcomes
MeSH Terms: conditions — Soft Tissue Injuries; Arthritis, Gouty; Fractures, Bone; Renal Colic; Dysmenorrhea; Agnosia; Sprains and Strains; Kidney Calculi; Emergencies

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- NSAID only: Subjects have their pain treated post-ED care with NSAID medication alone
- Opioid only: Subjects have their pain treated post-ED care with opioid medication alone
- NSAID + Opioid: Subjects have their pain treated post-ED care with NSAID medication and opioid as PRN rescue analgesia

SUMMARY:
Study aims to assess patient-recorded outcomes of pain control medications prescribed in the ER after visits for specific painful injuries/illnesses.

DETAILED DESCRIPTION:
Multicenter, observational, prospective, out-of-hospital registry collecting clinical, satisfaction, quality of life, and healthcare resource utilization from subjects discharged after ED care for a specific acute pain syndrome with a clinician-determined analgesic regimen. Subjects are stratified by diagnosis and by regimen based on the treating clinician's judgment. The registry study is independent of ED care and clinician's decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will meet the following criteria:

  1. Eligible diagnoses:

     musculoskeletal etiologies: acute extremity fractures sprains/strains acute gouty arthritis visceral etiologies: renal colic dysmenorrhea
  2. Age GTE 18 years;
  3. Decision to discharge from ED to community already made;
  4. Decision to give SPRIX, opioid, OR SPRIX + opioid rescue already made;
  5. Treating clinician deems patient appropriate for continued analgesic management as an outpatient for the next 3-5 days;
  6. Patient has ready touch-tone (mobile or land line) telephone access, provides number (and back-up number, if possible) and agrees (verbal or written consent as mandated by site) to answer and comply with brief IVR questionnaires daily for next 4 days.

Exclusion Criteria:

* Eligible subjects will meet none of the following criteria:

  1. Patient admitted or placed on observation status from ED;
  2. Patient unwilling or unable to comply with telephonic follow-up;
  3. Fracture that requires surgical repair (even if at a later date);
  4. Patient has diagnosis of any chronic pain syndrome;
  5. Patient already routinely takes NSAID or opioid agent;
  6. Treating clinician has reasonable suspicion of drug-seeking behavior or noncompliance;
  7. Nasal abnormality or illness that could affect the absorption of intranasal medication (such as: nasal discharge, rhinitis, acute upper respiratory infection, acute epistaxis, nasal polyp, nasal tumor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: at least 800 patients with specific musculoskeletal or visceral pain syndrome
Sampling Method: Non-Probability Sample
Enrollment: 843 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Clinical Outcomes of pain control measures | 5 days
  1. Change in pain score over follow-up interval;
  2. Healthcare resource utilization during follow-up interval;
  3. Patient satisfaction with therapy;
  4. Return to work in employed cohort.

SECONDARY OUTCOMES:
Satisfaction and Economic Outcomes | 5 days
  1. Effectiveness of work upon return;
  2. Relative adverse effect profiles of three treatment regimens;
  3. Compliance with therapy;
  4. QOL at conclusion of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Charles V Pollack, MD, Principal Investigator — University of Pennsylvania; Knox Todd, MD, Study Director — MD Anderson; Debra Diercks, MD, Study Director — UC Davis; Sharon Mace, MD, Study Director — The Cleveland Clinic; Stephen Thomas, MD, Study Director — Univ Oklahoma
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - LSU Medical Center, New Orleans, Louisiana
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma HSC, Tulsa, Oklahoma
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Ben Taub General Hospital, Houston, Texas
  - University of Texas HSC at Houston, Houston, Texas